CLINICAL TRIAL: NCT04696536
Title: Pilot Study: Twelve Week Clinical Efficacy of Supervised Mouth Rinse and Flossing: Effect on Plaque and Gingivitis
Brief Title: A Twelve Week Study of Supervised Mouth Rinse and Flossing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CCSORC000708; CCSORC000708 (Other: Johnson & Johnson Consumer Inc. (J&JCI))
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-04

CONDITIONS: Healthy
MeSH Terms: interventions — American Dental Association; Ethanol; Mouthwashes

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: Listerine Cool Mint Mouth Rinse (Marketed product) (Experimental): Participants will receive Alcohol-containing Essential Oil (AEO) containing mouth rinse (Listerine Cool Mint, marketed) orally for 12 weeks. Participant will brush their teeth and rinse once daily under supervision during the week (five days) for 30 seconds with 20 milliliter (mL) of mouth rinse and brush their teeth and rinse a second time each day during the week at home. During the weekends, participants will brush twice daily in their usual manner, following rinsing with their assigned mouth rinse, unsupervised at home.
  Interventions: Other: Colgate Cavity Protection Toothpaste; Other: American Dental Association (ADA) Referenced Toothbrush; Other: Alcohol-containing Essential Oil (AEO) Mouth Rinse (Listerine Cool Mint, marketed)
- Group 2: Negative Control (5 Percent (%) Hydroalcohol Mouth Rinse) (Experimental): Participants will receive negative control mouth rinse (5% Hydroalcohol mouth rinse) orally for 12 weeks. Participant will brush their teeth and rinse once daily under supervision during the week (five days) for 30 seconds with 20 milliliter (mL) of mouth rinse and brush their teeth and rinse a second time each day during the week at home. During the weekends, participants will brush twice daily in their usual manner, following rinsing with their assigned mouth rinse, unsupervised at home.
  Interventions: Other: Colgate Cavity Protection Toothpaste; Other: American Dental Association (ADA) Referenced Toothbrush; Other: 5% Hydroalcohol Mouth Rinse
- Group 3: Flossing Performed by Dental Hygienist (Experimental): Participants will brush their teeth and then undergo instructions on flossing technique using reach dental floss orally for 12 Weeks. Dental hygienist will floss participant's teeth at the site once daily during the week (five days). The second brushing will be done unsupervised at home. The remaining weekend days flossing and brushing will be done unsupervised at home.
  Interventions: Other: Colgate Cavity Protection Toothpaste; Other: American Dental Association (ADA) Referenced Toothbrush; Other: REACH Dental Floss
- Group 4: Flossing under Supervision (Experimental): Participants will brush their teeth and then undergo instructions on flossing technique using reach dental floss orally for 12 Weeks. Participants floss their teeth under supervision at the site once daily during the week (five days). The second brushing will be done unsupervised at home. The remaining weekend days flossing and brushing will be done unsupervised at home.
  Interventions: Other: Colgate Cavity Protection Toothpaste; Other: American Dental Association (ADA) Referenced Toothbrush; Other: REACH Dental Floss

INTERVENTIONS:
Other: Colgate Cavity Protection Toothpaste — Participants will use Colgate cavity protection toothpaste for brushing teeth twice daily.
Other: American Dental Association (ADA) Referenced Toothbrush — Participants will brush teeth at least one minute with provided toothbrush twice daily.
Other: 5% Hydroalcohol Mouth Rinse — Participants use 20 mL of 5% Hydroalcohol mouth rinse as negative control for 30 sec twice a day after brushing.
  Arms: Group 2: Negative Control (5 Percent (%) Hydroalcohol Mouth Rinse)
Other: REACH Dental Floss — Participants after brushing, rinse mouth with water and floss using Reach dental floss once a day.
  Arms: Group 3: Flossing Performed by Dental Hygienist; Group 4: Flossing under Supervision
Other: Alcohol-containing Essential Oil (AEO) Mouth Rinse (Listerine Cool Mint, marketed) — Participants after brushing, rinse with 20mL of the AEO mouth rinse for 30 seconds twice a day.
  Arms: Group 1: Listerine Cool Mint Mouth Rinse (Marketed product)

SUMMARY:
The purpose of this study is to evaluate the efficacy of twice daily alcohol containing essential oil mouth rinse and brushing versus dental flossing and brushing under once daily supervision for the prevention and reduction of plaque and gingivitis.

ELIGIBILITY:
Inclusion criteria:

* Able to comprehend and follow the requirements and restrictions of the study (including willingness to use the assigned study products according to instructions, availability on scheduled visit dates and likeliness of completing the clinical study) based upon research site personnel's assessment
* Able to attend once daily session during weekdays for flossing and rinsing occurring on site
* Evidence of a personally signed and dated informed consent document indicating the subject (or legally acceptable representative) has been informed of all pertinent aspects of the trial
* Able to read and understand the local language (participants capable of reading the documents)
* Adequate oral hygiene (that is brush teeth daily and exhibit no signs or oral neglect)
* A minimum of 20 natural teeth with scorable facial and lingual surfaces. Teeth that are grossly carious, extensively restored, orthodontically banded, abutments, exhibiting severe generalized cervical and/or enamel abrasion, or third molars will not be included in the tooth count
* A minimum of 10 bleeding sites based on the BI
* Absence of advanced periodontitis based on a clinical examination at Baseline and discretion of the dental examiner

Exclusion criteria:

* History of significant adverse effects, including sensitivities or suspected allergies, following use of oral hygiene products such as toothpastes, mouth rinses and red food dye
* Dental prophylaxis within four weeks prior to Screening/Baseline visit
* History of medical conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures
* Antibiotic, anti-inflammatory or anticoagulant therapy during the study or within the one month prior to the Baseline exam. Intermittent use of certain anti-inflammatory medication is acceptable at the discretion of the Investigator
* Use of chemotherapeutic anti-plaque/anti-gingivitis products such as triclosan, essential oils, cetylpyridinium chloride, stannous fluoride or chlorhexidine containing mouth rinses within the two weeks prior to Baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Interproximal Mean Turesky Plaque Index (TPI) Score After 12 Weeks of Product use | 12 Weeks
  Plaque area will be assessed using the Turesky Modification of the Quigley- Hein Plaque Index, on six surfaces (disto-buccal, mid-buccal, mesio-buccal and disto-lingual, mid-lingual, and mesio-lingual) of all scorable teeth, following disclosing: 0 - No plaque; 1 - Separate flecks or discontinuous band of plaque at the gingival (cervical0 margin); 2- Thin (up to 1 millimeter), continuous band of plaque at the gingival margin; 3 - Band of plaque wider than 1 mm but less than 1/3 of surface; 4 - Plaque covering 1/3, but less than 2/3 of surface; 5 - Plaque covering 2/3 or more of a surface.
Interproximal Mean Modified Gingival Index (MGI) Score After 12 Weeks of Product use | 12 Weeks
  Gingivitis will be assessed using Modified Gingival Index on the buccal and lingual marginal gingivae and interdental papillae of all scorable teeth: 0- Normal (absence of inflammation); 1- Mild inflammation (slight change in color, little change in texture) of any portion of the entire gingival unit; 2- Mild inflammation of the entire gingival unit; 3- Moderate inflammation (moderate glazing, redness, edema, and/or hypertrophy) of the gingival unit; 4- Severe inflammation (marked redness and edema/hypertrophy, spontaneous bleeding, or ulceration) of the gingival unit.

SECONDARY OUTCOMES:
Interproximal Mean Turesky Plaque Index (TPI) Score After 4 Weeks of Product use | 4 Weeks
  Plaque area will be assessed using the Turesky Modification of the Quigley- Hein Plaque Index, on six surfaces (disto-buccal, mid-buccal, mesio-buccal and disto-lingual, mid-lingual, and mesio-lingual) of all scorable teeth, following disclosing: 0 - No plaque; 1 - Separate flecks or discontinuous band of plaque at the gingival (cervical0 margin); 2- Thin (up to 1 millimeter), continuous band of plaque at the gingival margin; 3 - Band of plaque wider than 1 mm but less than 1/3 of surface; 4 - Plaque covering 1/3, but less than 2/3 of surface; 5 - Plaque covering 2/3 or more of a surface.
Interproximal Mean Modified Gingival Index (MGI) Score After 4 Weeks of Product use | 4 Weeks
  Gingivitis will be assessed using Modified Gingival Index on the buccal and lingual marginal gingivae and interdental papillae of all scorable teeth: 0- Normal (absence of inflammation); 1- Mild inflammation (slight change in color, little change in texture) of any portion of the entire gingival unit; 2- Mild inflammation of the entire gingival unit; 3- Moderate inflammation (moderate glazing, redness, edema, and/or hypertrophy) of the gingival unit; 4- Severe inflammation (marked redness and edema/hypertrophy, spontaneous bleeding, or ulceration) of the gingival unit.
Whole-mouth Mean Turesky Plaque Index (TPI) Score After 4 Weeks and 12 Weeks of Product use | 4 Weeks and 12 Weeks
  Plaque area will be assessed using the Turesky Modification of the Quigley- Hein Plaque Index, on six surfaces (disto-buccal, mid-buccal, mesio-buccal and disto-lingual, mid-lingual, and mesio-lingual) of all scorable teeth, following disclosing: 0 - No plaque; 1 - Separate flecks or discontinuous band of plaque at the gingival (cervical0 margin); 2- Thin (up to 1 millimeter), continuous band of plaque at the gingival margin; 3 - Band of plaque wider than 1 mm but less than 1/3 of surface; 4 - Plaque covering 1/3, but less than 2/3 of surface; 5 - Plaque covering 2/3 or more of a surface.
Whole-mouth Mean Modified Gingival Index (MGI) Score After 4 Weeks and 12 Weeks of Product use | 4 Weeks and 12 Weeks
  Gingivitis will be assessed using Modified Gingival Index on the buccal and lingual marginal gingivae and interdental papillae of all scorable teeth: 0- Normal (absence of inflammation); 1- Mild inflammation (slight change in color, little change in texture) of any portion of the entire gingival unit; 2- Mild inflammation of the entire gingival unit; 3- Moderate inflammation (moderate glazing, redness, edema, and/or hypertrophy) of the gingival unit; 4- Severe inflammation (marked redness and edema/hypertrophy, spontaneous bleeding, or ulceration) of the gingival unit.
Whole-mouth and Interproximal Mean Bleeding Index (BI) After 4 and 12 Weeks of Product use | 4 Weeks and 12 Weeks
  Bleeding will be assessed according to the Gingival Bleeding Index. A periodontal probe with a 0.5 mm diameter tip will be inserted into the gingival crevice and swept from distal to mesial around the tooth at an angle of approximately 60 degree, while in contact with the sulcular epithelium. Each of 4 gingival areas (distobuccal, mid-buccal, mid-lingual, and mesiolingual) around each tooth will be assessed. After approximately 30 seconds, bleeding at each gingival unit will be recorded according to the following scale: 0- Absence of bleeding after 30 seconds; 1- Bleeding after 30 seconds; 2- Immediate bleeding.
Whole-mouth and Interproximal Percent Bleeding Sites, Based on the BI Score After 4 and 12 Weeks of Product use | 4 Weeks and 12 Weeks
  Bleeding will be assessed according to the Gingival Bleeding Index. A periodontal probe with a 0.5 mm diameter tip will be inserted into the gingival crevice and swept from distal to mesial around the tooth at an angle of approximately 60 degree, while in contact with the sulcular epithelium. Each of 4 gingival areas (distobuccal, mid-buccal, mid-lingual, and mesiolingual) around each tooth will be assessed. After approximately 30 seconds, bleeding at each gingival unit will be recorded according to the following scale: 0- Absence of bleeding after 30 seconds; 1- Bleeding after 30 seconds; 2- Immediate bleeding.
Interproximal of the Proximal Marginal Plaque Index Score After 4 and 12 Weeks | 4 Weeks and 12 Weeks
  Interproximal Plaque area will be assessed using the PMI on the facial and lingual surfaces. Distal proximal and mesial proximal will be assessed on all teeth including the distal of the second molar using the following scoring system: 0- No plaque; 1 - Separate flecks of plaque covering less than 1/3 of the area; 2 - Discrete areas or bands of plaque covering less than 1/3 of the area; 3 - Plaque covering 1/3 of the area; 4 - Plaque covering more than 1/3 but less than 2/3 of the area; 5 - Plaque covering 2/3 or more of the area.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Milleman, DDS, Principal Investigator — Salus Research, Inc.
Locations (1):
- Salus Research, Inc., Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

REFERENCES:
- [Background] Bauroth K, Charles CH, Mankodi SM, Simmons K, Zhao Q, Kumar LD. The efficacy of an essential oil antiseptic mouthrinse vs. dental floss in controlling interproximal gingivitis: a comparative study. J Am Dent Assoc. 2003 Mar;134(3):359-65. doi: 10.14219/jada.archive.2003.0167. PMID 12699051
- [Background] Marsh PD. Controlling the oral biofilm with antimicrobials. J Dent. 2010 Jun;38 Suppl 1:S11-5. doi: 10.1016/S0300-5712(10)70005-1. PMID 20621238
- [Background] Sharma NC, Charles CH, Qaqish JG, Galustians HJ, Zhao Q, Kumar LD. Comparative effectiveness of an essential oil mouthrinse and dental floss in controlling interproximal gingivitis and plaque. Am J Dent. 2002 Dec;15(6):351-5. PMID 12691269
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CCSORC000708&attachmentIdentifier=181f1518-6d87-432c-8c92-ce12f07a453e&fileName=CCSORC00708___CSR_Synopsis_for_ClinTrials___24_Feb_2021.gov___Redacted_Redacted_PDF_A.pdf&versionIdentifier=